CLINICAL TRIAL: NCT03189992
Title: Study of "Same TCM Syndrome for Different Diseases" and "Same Treatment for Different Diseases" of Primary Hepatocellular Carcinoma and Colorectal Cancer Under the Perspective of System Science
Brief Title: Study of TCM Syndrome of Hepatocellular Carcinoma and Colorectal Cancer Based on System Science
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ShanghaiUTCM
Record Dates: First submitted 2017-06-04; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-03

CONDITIONS: Malignant Tumor of Small Intestine Metastatic to Liver
MeSH Terms: interventions — cinobufotalin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CC-GSYXZ (Experimental): Colon cancer with Chinese medicine syndrome Yin deficiency of liver and kidney and spleen deficiency.Intervented by Bushen-Jianpi Dedoction and cinobufotalin injection
  Interventions: Drug: Bushen-Jianpi Dedoction; Drug: cinobufotalin injection
- CC-WZ (Placebo Comparator): Colon cancer with none Chinese medicine syndrome.Intervented by cinobufotalin injection
  Interventions: Drug: cinobufotalin injection
- HCC-GSYXZ (Experimental): Hepatoma cancer with Chinese medicine syndrome Yin deficiency of liver and kidney and spleen deficiency.Intervented by Bushen-Jianpi Dedoction and cinobufotalin injection.
  Interventions: Drug: Bushen-Jianpi Dedoction; Drug: cinobufotalin injection
- HCC-WZ (Placebo Comparator): Hepatoma cancer with none Chinese medicine syndrome.Intervented by cinobufotalin injection
  Interventions: Drug: cinobufotalin injection

INTERVENTIONS:
Drug: Bushen-Jianpi Dedoction — A traditional chinese medicine prescription
  Other Names: BSJPD
  Arms: CC-GSYXZ; HCC-GSYXZ
Drug: cinobufotalin injection — an effective Chinese preparation to treat malignant tumor.
  Other Names: CI

SUMMARY:
Traditional Chinese medicine (TCM) syndrome is a core foundation of disease knowledge, clinical diagnosis and treatment and curative effect evaluation in TCM. "Same TCM Syndrome for Different Diseases" and "Same Treatment for Different Diseases" is one of the characteristics of TCM syndrome differentiation and treatment.

This study is the "TCM disease syndrome combination" research baced on principles and methods of system biology, which is through acquisition of primary hepatocellular carcinoma (HCC) and colorectal cancer patients with TCM syndrome information, detection of clinical indicators and genomic, proteomic, and metabolites changes, analyzing the correlation between TCM syndromes and biological information, and revealing its biological material characteristics and the molecular mechanisms of "Same TCM Syndrome for Different Diseases";Developing and implementing the program of TCM syndrome differentiation and treatment for HCC and colorectal cancer to evaluate the efficacy of TCM syndrome based-treatment of HCC and colorectal cancer with TCM syndrom scores, clinical and systems biological indicators, quality of life and survival rate, and to revealing the mechanism of the "Same Treatment for Different Diseases".

DETAILED DESCRIPTION:
Traditional Chinese medicine (TCM) syndrome is a core foundation of disease knowledge, clinical diagnosis and treatment and curative effect evaluation in TCM. "Same TCM Syndrome for Different Diseases" and "Same Treatment for Different Diseases" is one of the characteristics of TCM syndrome differentiation and treatment.

In this study, the investigators adopted the transcriptome analysis, proteome analysis and metabolic diversity analysis of the patients with different syndromes of liver cancer and colorectal cancer, and integrate omics information, combining macro and micro methods to screen biomarkers of syndromes

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of primary liver cancer (HCC) and colorectal cancer after surgery.
2. Liver cancer and colorectal cancer liver and kidney yin deficiency and spleen qi deficiency syndrome diagnosis standard : Yin deficiency of liver and kidney and spleen qi deficiency syndrome see hypochondriac pain, waist and knee Limp, fever, night sweats, dry mouth and throat, fatigue, anorexia, abdominal distension after eating more, red or pale tongue, less moss or Light peel, pulse fine.

Exclusion Criteria:

(1) there is a serious heart, kidney, and other diseases of the hematopoietic system effect of drug evaluation factors; (2)Mental disorders (3)Digestive tract obstruction; (4) poor compliance.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Complete patient recruitment | 24 months
  Complete transcriptome microarray detection

CONTACTS AND LOCATIONS:
Overall Officials: shi bing su, PhD, Principal Investigator — Shuguang Hospital affiliated with Shanghai University of TCM
Locations (1):
- Shang Hai TCM University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang J, Hu Y, Zhao K, Fan J, Zhu J, Li Q, Chen Q, Lu Y. Comprehensive Analysis of the Expression of Cell Adhesion Molecules Genes in Hepatocellular Carcinoma and their Prognosis, and Biological Significance. Front Biosci (Landmark Ed). 2024 Feb 21;29(2):76. doi: 10.31083/j.fbl2902076. PMID 38420809
- [Derived] Chen J, Chen QL, Wang WH, Chen XL, Hu XQ, Liang ZQ, Cao YB, Cao YM, Su SB. Prognostic and predictive values of CXCL10 in colorectal cancer. Clin Transl Oncol. 2020 Sep;22(9):1548-1564. doi: 10.1007/s12094-020-02299-6. Epub 2020 Feb 3. PMID 32016676
- [Derived] Lu Y, Fang Z, Zeng T, Li M, Chen Q, Zhang H, Zhou Q, Hu Y, Chen L, Su S. Chronic hepatitis B: dynamic change in Traditional Chinese Medicine syndrome by dynamic network biomarkers. Chin Med. 2019 Nov 21;14:52. doi: 10.1186/s13020-019-0275-4. eCollection 2019. PMID 31768187